CLINICAL TRIAL: NCT01878864
Title: Effect of Local Anesthesia in Patients With Marginal Periodontitis Undergoing Scaling and Root Planning
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too slow patient inclusion and superior effect of the injection
Sponsor: Ove Andersen (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, MD, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OC004PDS; 2012-003430-16 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-06-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Pain and Discomfort During Scaling and Root Planning of Patients With; Periodontitis
Keywords: Pain, Discomfort, Periodontitis, Scaling and Root Planning, Visual Analogue Scale, McGills Pain Questionnaire
MeSH Terms: conditions — Pain; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine lozenge (Experimental): Single dose administration of a 25 mg bupivacaine lozenge before the scaling and root planning was performed.
  Interventions: Drug: Bupivacaine lozenge
- Lidocaine-adrenalin injection (Active Comparator): Xyloplyin Dental Adrenalin (20 mg/ml lidocaine, 12.5 microgram/ml adrenaline). Frequency and duration of injections was decided by the dentist preforming the scaling and root planning.
  Interventions: Drug: Lidocaine-adrenalin injection

INTERVENTIONS:
Drug: Bupivacaine lozenge
  Arms: Bupivacaine lozenge
Drug: Lidocaine-adrenalin injection
  Arms: Lidocaine-adrenalin injection

SUMMARY:
A randomised cross-over study comparing two methods of local anaesthesia for patients diagnosed with periodontitis undergoing scaling and root planning. 40 patients will be included in the study, which aims to demonstrate that the effect of a bupivacaine lozenge is non-inferior to lidocaine-adrenalin injections.

DETAILED DESCRIPTION:
40 periodontitis patients undergoing scaling and root planning (SRP) will be randomised to receive local anaesthesia by either a bupivacaine lozenge or lidocaine-adrenalin injection at their first visit. At the following visit, the patients will receive the opposite treatment.

At each visit the patient will evaluate pain before, during and after SRP by:

* Visual Analog Scale (VAS) 0-10 where 0 = no pain, 10 = extreme pain.
* McGills Pain Questionnaire (MPQ), which gives a qualitative pain profile.

At each visit the patient will evaluate discomfort before, during and after the SRP by:

- Visual Analog Scale (VAS) 0-10 where 0 = no discomfort, 10 = extreme discomfort.

Additionally the patient assesses the comfort of administration of the two local anaesthesia as well as the taste of the bupivacaine lozenge. The investigator also evaluates the scaling procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having, respectively periodontitis marginalis adulta progressiva lenta and periodontitis marginalis adulta progressiva rapid in the hygiene phase, where depurations are repeated within a short timeframe
* Age between 18 and 80 years
* Ability to speak, read and understand danish
* Ability to give oral and written consent

Exclusion Criteria:

* Known allergy to bupivacaine or other local anaesthetics of the amide type
* Other gingival infections (eg lichen planus)
* Pregnancy -if in doubt a pregnancy test will be made
* Breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate a non-inferior effect on pain and discomfort during scaling and root planning by a bupivacaine lozenge in comparison to lidocaine-adrenalin injections. | Day 1
  Pain and discomfort are measured immediately after the scaling and root planning procedure
  Level of pain:
  -Visual Analog Scale (VAS) 0-10 where 0 = no pain, 10 = extreme pain
To demonstrate a non-inferior effect on pain and discomfort during scaling and root planning by a bupivacaine lozenge in comparison to lidocaine-adrenalin injections. | Day 1
  Pain and discomfort are measured immediately after the scaling and root planning procedure
  Level of discomfort:
  -Visual Analog Scale (VAS) 0-10 where 0 = no discomfort, 10 = extreme discomfort

SECONDARY OUTCOMES:
Investigator evaluation of the scaling procedure | Day 1
  After the scaling and root planning the investigator evaluates the scaling procedure by a questionnaire
Patient assessment of the two pharmaceutical formulations | Day 1
  After the scaling procedure the patient assesses the two pharmaceutical formulations by a questionnaire
To demonstrate a non-inferior effect on pain and discomfort during scaling and root planning by a bupivacaine lozenge in comparison to lidocaine-adrenalin injections. | Daiy 1
  Pain and discomfort are measured immediately after the scaling and root planning procedure
  Level of pain:
  -McGills Pain Questionnaire (MPQ), which gives a qualitative pain profile

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, MD, Study Director — Hvidovre UH
Locations (3):
- Denmark (3):
  - Tandlægerne Vimmelskaftet, Copenhagen K
  - Frederiksberg Tandlægerne, Frederiksberg
  - Tandlægepraksis ved Jonna Bork, Hvidovre